CLINICAL TRIAL: NCT01480973
Title: MRI Assessment of Post-Radiation Change Following Stereotactic Body RT for Non-Small Cell Lung Cancer: A Pilot Study
Brief Title: Stereotactic Body Radiotherapy (RT) for Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 11-0079-CE
Record Dates: First submitted 2011-08-16; First posted 2011-11-29 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

ARMS (1):
- MRI post lung SBRT (Experimental): Feasibility of MRI to differentiate between benign and malignant changes seen after lung SBRT.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — SBRT involves highly precise delivery of very high dose Radiotherapy (RT) over a very few fractions (hypofractionation) to accurately delineated, size-restricted malignant targets in which motion has been accounted for during the delivery process. SBRT administration achieves avoidance of normal tissue exposure to radiation during the planning process, by providing for sharp fall-off dose gradients outside the target.

SUMMARY:
NSCLC is the leading cause of cancer mortality in North America, accounting for nearly 30% of all cancer deaths. The standard treatment for patients with early-stage non-small-cell lung cancer (NSCLC) is surgical resection of the involved lobe/lung. However, many patients are unable to undergo such a major surgery due to medical illness, and an emerging standard-of-care for these patients stereotactic-body radiation therapy (SBRT).

SBRT involves highly precise delivery of very high dose Radiotherapy (RT) over a very few fractions (hypofractionation) to accurately describe, size-restricted malignant targets in which motion has been accounted for during the delivery process. SBRT administration achieves avoidance of normal tissue exposure to radiation during the planning process, by providing for sharp fall-off dose gradients outside the target.

ELIGIBILITY:
Inclusion Criteria:

* Must have been treated at University of Health Network with SBRT for an early-stage NSCLC (T1N0M0; T2N0M0; or T3N0M0 chest wall primary tumours only).
* On follow-up thoracic CT scans, patients must have changes in the previously targeted lung parenchyma that fit into one of the following three patterns: - Changes that on CT and clinical grounds are felt to be related to fibrosis
* Changes that on CT and clinical grounds are suspicious for recurrence
* Equivocal changes (uncertain whether the changes represent fibrosis or recurrence)
* Must be greater than 18 years in age
* Must be able to attend regular follow-up including radiologic investigations and clinical visits
* Written informed consent

Exclusion Criteria:

* Standard contraindications to MRI study (e.g. ferromagnetic prosthesis, pacemaker/implanted defibrillator, metallic implant in eye, severe claustrophobia, etc…)
* Contraindications to Gadolinium contrast-agent. May include a history of allergic reaction to following previous administration of gadolinium or poor renal function (calculated creatinine clearance < 30 mL/min).
* Patients with surgical resection of the treated portion of lung following their SBRT, although surgical resection of other parts of the lung is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2017-07 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Optimal MRI parameters and sequences to characterize lung changes observed after SBRT for early-stage NSCLC. | 2 years
  MRI pulse sequence settings
MRI characteristics of benign (fibrosis), malignant (recurrence), and indeterminate lung changes observed after SBRT for early-stage NSCLC. | 2 years
  MRI tissue contrast

SECONDARY OUTCOMES:
Reliability and reproducibility of thoracic MRI to distinguish between benign (fibrosis), malignant (recurrence), and indeterminate lung changes following SBRT for early-stage NSCLC. | 2 years
  Sensitivity, specificity, positive and negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: John Cho, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, University Health Network, Toronto, Ontario, Canada